CLINICAL TRIAL: NCT04049188
Title: Impact of Access to Single-Fraction Palliative Radiation Therapy in Cancer Patients Enrolled in Hospice
Brief Title: Access to Single-Fraction Palliative Radiation Therapy in Cancer Patients Enrolled in Hospice
Acronym: SFPRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Care Partners (Other)
Collaborators: OHSU Knight Cancer Institute (Other); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00019460; 20181015 (Other Grant/Funding Number: Knight Cancer Institute - Community Partnership Program)
Record Dates: First submitted 2019-03-05; First posted 2019-08-08 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Cancer Metastatic
Keywords: Cancer Patients Hospice Care; Palliative Radiation Therapy
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Fraction Palliative RT (Experimental): Single-Fraction Palliative Radiation Therapy Adminstration
  Interventions: Radiation: Single-Fraction Palliative Radiation Therapy

INTERVENTIONS:
Radiation: Single-Fraction Palliative Radiation Therapy — All subjects will be undergo single-fraction palliative radiation therapy who have cancer and associated bone metastases and symptomatic bone pain.

SUMMARY:
Feasibility study to report on the impact of ACCESS of single-fraction radiation therapy on cancer patients with bone metastases enrolled in hospice care.

DETAILED DESCRIPTION:
Hospice care for terminally ill patients with metastatic cancer improves quality of life, pain control, and potentially also survival when patients are enrolled early.1-3 However, hospice programs are often seen by patients and their caregivers as the last resort after exhaustion of all effective treatment options. The need to revoke active treatment (for all hospice patients with cancer outside of the VA system) discourages hospice enrollment.

This study aims to understand and analyze barriers to access specifically for short course palliative radiation therapy in cancer patients enrolled in hospice.

ELIGIBILITY:
Inclusion Criteria:

* Solid Tumor Malignancies and Multiple Myeloma with Bone Metastases and Associated Bone Pain Enrolled in Hospice

Exclusion Criteria:

* Decisionally-Impaired Subjects, Pregnant Women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Opioid Use for Pain Management | Through study completion, an average of 1 year
  Opioid Dosage (mg/day)

SECONDARY OUTCOMES:
Improved Quality of Life Measures | During study completion
  Questionnaires using Herth Hope Index, Timed Up and Go, and Edmonton Symptom Assessment Scale
Improved Activities of Daily Living | During study completion
  Questionnaires using Hearth Hope Index, Timed Up and Go, and Edmonton Symptom Assessment Scale

CONTACTS AND LOCATIONS:
Locations (1):
- CarePartners, Hillsboro, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided